CLINICAL TRIAL: NCT03937622
Title: Northern Survey on Therapeutic Oxygen Prescription
Acronym: NONSTOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Pneumo-O2
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Oxygen Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 17 items questionaire — This is a prospective multicenter observational trial. Included patients and attending physician complete a standardised questionnaire.

SUMMARY:
This is a prospective multicenter observational trial. Included patients and attending physician complete a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lung disease, age > 18 years
* Established domiciliary LTOT > 4 weeks
* Scheduled for control of oxygen therapy with arterial/capillary

Exclusion Criteria:

* No informed consent
* Pulmonary exacerbation within the last 2 weeks
* Signs of heart failure (edema, congestion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the Inclusion criteria and not the exclusion criteria at 3 Centers in nothern Germany
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Validation of indication of Long-term Oxygen therapy (LTOT) | 12 month
  Aim of this study is to observe the real-world handling with longterm Oxygen treatment in northern Germany

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, Prof. Dr. med., Principal Investigator — Hannover Medical School
Locations (2):
- Germany (2):
  - Dep. Respiratory Medicine, Hannover Medical School, Hanover
  - Department of Respiratory Medicine, Medizinische Hochschule Hannover, Hanover

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participants data